CLINICAL TRIAL: NCT01997606
Title: Cross-over Study of the Impact of Purotex Covers on the Concentration of House Dust Mite Allergen in Bedding and the Quality of Life in Patients With Allergic Rhinitis to House Dust Mite.
Brief Title: House Dust Mite Allergen Reduction in Bedding: Purotex Impregnated Covers of Bekaert Textiles
Acronym: Purotex covers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Bekaert textiles NV Waregem (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012/398
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purotex (Experimental): use of Purotex treated bedding covers
  Interventions: Other: use of Purotex treated bedding covers
- Placebo (Placebo Comparator): no use of Purotex treated bedding covers
  Interventions: Other: placebo

INTERVENTIONS:
Other: use of Purotex treated bedding covers — Purotex is a textile treatment that uses five 100% natural bacteria or probiotics, selected for their ability to clean up house dust mite allergen along with other allergen types. The active probiotics are placed inside of millions of capsules and are introduced during the textile production. These human friendly bacteria remain non-active until friction force is created between the mattress/pillow and the sleeper's body. Under the friction force a small part of the capsules is opened and probiotics become active. They saturate the bacterial capacity of the textile and by doing so, reduce the risk of dust mite allergen development and growth of molds and harmful bacteria. The patients will apply the covers around their mattress and around their pillow. On top of these covers the patients will apply their own fitted sheet and pillowcase (which they will change every 4 weeks).
  Arms: Purotex
Other: placebo
  Arms: Placebo

SUMMARY:
Product information:

Purotex is a textile treatment that uses five 100% natural bacteria or probiotics, selected for their ability to clean up house dust mite allergen along with other allergen types.

Study design:

* Placebo-controlled: the effect of the Purotex impregnated mattress and pillow covers will be compared to untreated, classical bedding covers (placebo).
* Cross-over design: There will be 2 'treatment' arms. One arm (Arm 1) in which the subjects will first use the Purotex impregnated covers (Set A=Purotex) during 2 months (=period A) and, after a wash out period of 1 month, the untreated covers (set B=placebo) during 2 months (=period B). In the second arm (Arm 2), the subjects will first use the untreated set (set A=placebo) and, after a wash out period the Purotex impregnated covers (set B=Purotex).
* Randomized: The subjects will be randomly assigned to one of the 2 treatment arms.
* Double blind: both the subjects and the investigators will not know to which treatment arm the subjects are assigned.

Study hypothesis:

We want to investigate:

* if there is a reduced concentration of HDM allergen in Purotex covers compared to untreated covers in real life
* if patients with allergic rhinitis to house dust mite use the Purotex covers, they experience an improvement of their quality of life and sleep, and an improvement of their allergic symptoms and global discomfort

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing to give/sign informed consent
* Subjects (male or female) must be at least 18 years old and maximum 65 years old at screening
* Clinical history of allergic rhinitis for at least 1 year
* Positive skin prick test for D. Pteronyssinus ± D. Farinae
* Positive nasal provocation test with the house-dust-mite allergen
* Specific IgE: Unicap positive to D. Pteronyssinus (d1) and D. Farinae (d2) (> 0.7U/ml)
* VAS score for global discomfort caused by nasal- or other allergic symptoms during the previous 4 weeks ≥ 5.
* The concentration of Der p1 in the dust collected from own bedding (mattress and pillow), measured by ELISA is above the detection limit (≥ 0.488 ng/ml).

Exclusion Criteria:

* Patients sensitized to animals should not be included if they are symptomatic upon exposure and regularly exposed to animals: positive SPT to pets and pets at home
* Patients with an allergy to tree pollen (symptoms during the season + positive skin prick test) should not be included
* Subject pregnant or lactating
* Completed allergen specific immunotherapy (SCIT or SLIT) with HDM within the last 5 years
* SCIT or SLIT during the study period
* Regular use of oral corticosteroids for exacerbations of asthma
* Daily use of oral corticosteroids
* Daily use of cyclosporine or other immunosuppressant drugs
* Regular use of antibiotics
* History of anaphylactic reaction to an allergen
* Severe general diseases (especially cardiopulmonary disease with reduced lung capacity)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in house dust mite allergen concentration | every two weeks, starting after randomisation untill completion of the study (5 months after randomisation)
  Concentration of house dust mite allergen in dust collected from the mattress and pillow covers will be measured by using ELISA During the study, the patients will collect dust every 2 weeks (for each cover their will be 5 time points with an interval of 2 weeks on which dust will be collected)

SECONDARY OUTCOMES:
Change in quality of life | every week during the course of the study (from baseline untill 5 months after)
  questionnaires: RQLQ, NRQLQ
change in quality of sleep | every week during the course of the study (from start till 5 months)
change in control of allergic rhinitis symptoms | every week during the course of the study (from baseline till month 5)
  questionnaire
change in global discomfort | every week during the course of the study (from baseline till month 5)
  global discomfort due to allergic symptoms and discomfort from specific symptoms questionnaire VAS
change in use of rescue medication | every week during the course of the study (from baseline till month 5)
  patients will fill out every week a questionnaire about the use of medication for their allergic rhinitis (and asthma)
change in discomfort during sleep | every week during the course of the study (from baseline till month 5)

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium